CLINICAL TRIAL: NCT00145379
Title: The Effect of Metformin in Overweight Patients With Dysregulated Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 006
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; insulin resistance; metformin; randomized, controlled study
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

ARMS (2):
- Metformin (Experimental)
  Interventions: Drug: Tablet Metformin 500 mg
- Placebo comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tablet Metformin 500 mg
  Arms: Metformin
Drug: Placebo
  Arms: Placebo comparator

SUMMARY:
Patients suffering from diabetes through many years have a risk of developing late diabetic complications including changes in eyes, kidney, vessels and nerves. Late complications can be postponed or avoided when assuring a good diabetes control, i.e. sensible diet, exercise, frequent blood glucose measurements and a good medical treatment.

Blood glucose regulation depends on two different factors i.e. the insulin need of the body and the amount of insulin in the body. The amount of insulin, in blood, is decided by the amount of insulin infused daily, whereas the insulin need depends on the patient's weight, physical activity and diet. Overweight type 2 diabetes patients have a large insulin need and especially this need is decisive for their development of diabetes. If these patients are treated with Metformin, blood glucose decreases and the result is an easier weight loss for the patient. Especially, when these patients take this drug, the development of late diabetic complications, especially arteriosclerosis, can be avoided or postponed.

Whether these favourable effects of Metformin are also present in type 1 diabetic patients remains to be fully clarified, but some studies have indicated that this is the case. This results in a better regulation of diabetes on a smaller insulin dose than the one given to the patients before.

Metformin probably takes effect by increasing the glucose uptake in muscles and by reducing the hepatic glucose production. The drug usually has no side-effects, but some patients do, however, suffer from abdominal pain, small tendency to nausea, loose defaecation and a metallic taste in the mouth. These side-effects are often temporary.

Project description

In total, 50 type 1 diabetic patients are offered to participate in the project. All are from the outpatient clinic at the Department of Endocrinology. The project lasts 7 months divided as follows:

1. An introductory period of one month introducing an optimisation of the insulin treatment
2. A 6 month period (in which neither the patients nor the treating doctor know which medication is given) with either T. Metformin treatment twice daily or T. Placebo (lime) twice daily together with the usual insulin treatment four times daily.

Choice of either T. Metformin or T. Placebo will be made by draw, and as stated above, the drug type will be unknown for both the patient and the treating doctor in order to make sure that the investigation is as objective as possible.

Throughout the examination period, the patients are asked to measure blood glucose four times daily, i.e. before main meals and before bed time. These values will be used for regulating the fasting insulin dose with help from the treating doctor, and for adjusting the daily insulin dose. During the first and the last two days of the examination period we will also ask the patients to measure blood glucose at 03h00 for two days. Those diurnal profiles will be included in the evaluation of the blood glucose control during the treatment period. Furthermore, the patients' blood pressures are determined during 24 hours before and after the 6 months' treatment period. This will be carried out automatically by means of a blood pressure cuff around the arm connected to a small apparatus registering the values during 24 hours. The apparatus can be taken home after installation at the outpatient clinic and can be carried around in a belt around the waist until next day where the apparatus will be dismantled.

At the first and the last of 5 outpatient visits, blood tests will be taken (for evaluation of the long-term blood glucose, kidney, liver, insulin and fat in blood) and nocturnal urine must be collected and disposed in order to evaluate protein secretion and thereby kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes mellitus treated with insulin 4 times daily.
* Age: 18-60 years
* Fertile women use adequate contraception, e.g. contraceptive pills
* C-peptide <300 pmol/L
* BMI >/= 25
* HbA1c >/=8%

Exclusion Criteria:

* Pregnant and patients planning to become pregnant during the investigation period
* Reduced eyesight
* Known kidney disease, s-creatinin >100
* Liver disease, Alat > 50
* Neuropathic patients diagnosed by clinical examination

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2003-03; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
HbA1c after the two intervention periods

SECONDARY OUTCOMES:
Insulin need, hypoglycaemia frequence, body weight, lipid profile, blood pressure after the two intervention periods

CONTACTS AND LOCATIONS:
Overall Officials: Iben Brock Jacobsen, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Diabetes Research Center, Odense, Funen, Denmark